CLINICAL TRIAL: NCT03617445
Title: Fecal Microbiota Transplantation for C. Difficile Infection in Solid Organ Transplant Recipients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study drug not available due to COVID-19 FDA restrictions
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-1056; A534265 (Other: UW Madison); SMPH/MEDICINE/INFECT DIS (Other: UW Madison); Protocol Version 8/24/2022 (Other: UW Madison); 1U01AI125053-01A1 (NIH)
Record Dates: First submitted 2018-07-27; First posted 2018-08-06 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Clostridium Difficile Infection Recurrence
MeSH Terms: interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Intervention Model Description: This is a phase 2, double blind, doubly placebo-controlled, randomized trial assessing the treatment effects of FMT compared to oral Vancomycin for recurrent CDI in solid organ transplant recipients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- FMT oral capsules/ oral vancomycin placebo (Active Comparator): FMT plus placebo vancomycin
  Interventions: Drug: FMT oral capsule; Drug: Oral Vancomycin placebo
- Placebo FMT capsules/ Active oral vancomycin (Active Comparator): Vancomycin plus FMT enema placebo
  Interventions: Drug: Oral Vancomycin; Drug: FMT oral placebo

INTERVENTIONS:
Drug: FMT oral capsule — FMT oral capsules, single dose of 5 capsules
  Other Names: MTP-101-C
  Arms: FMT oral capsules/ oral vancomycin placebo
Drug: Oral Vancomycin — Oral Vancomycin 125 mg capsules every 6 hours for 14 days, followed by 125 mg oral placebo every 12 hours for 7 days, followed by 125 mg oral placebo once daily for 7 days, followed by 125 mg oral placebo every 3 days for 14 days
  Other Names: vancomycin
  Arms: Placebo FMT capsules/ Active oral vancomycin
Drug: FMT oral placebo — Placebo oral capsules, single dose of 5 capsules
  Other Names: Placebo MTP-101-C
  Arms: Placebo FMT capsules/ Active oral vancomycin
Drug: Oral Vancomycin placebo — Placebo oral vancomycin capsules every 6 hours for 14 days, followed by 125 mg oral vancomycin every 12 hours for 7 days, followed by 125 mg oral vancomycin once daily for 7 days, followed by 125 mg oral vancomycin every 3 days for 14 days.
  Other Names: placebo
  Arms: FMT oral capsules/ oral vancomycin placebo

SUMMARY:
The objective is to examine the effect of Fecal Microbiota Transplantation (FMT) compared with vancomycin for cure of recurrent C. diff infection (CDI) in solid organ transplant (SOT) recipients in a randomized, controlled clinical trial.

DETAILED DESCRIPTION:
Clostridium difficile (C.difficile) is a pathogen of major public health importance, especially in individuals with comorbid conditions such as solid organ transplantation (SOT). The incidence and adverse outcomes of CDI are greatly amplified in the setting of SOT, due to healthcare exposure, antibiotic use and immunosuppression, all of which are ubiquitous in SOT recipients. There are currently no effective treatment options to achieve a sustained cure of recurrent CDI and prevent further recurrence in SOT recipients. A novel approach that has recently gained attention is restoration of the CDI impaired gut microbiome by instillation of stool from a healthy donor into the intestine of a CDI patient. This treatment, called Fecal Microbiota Transplantation (FMT) has been found in non-comparative studies to reduce CDI recurrence dramatically with a reported efficacy of over 95%, however its efficacy in SOT recipients has not been studied and cannot be extrapolated from results in the non-SOT population because SOT recipients are a unique study population due to profound immunosuppression, frequent antibiotic use and frequent opportunities for exposure to CDI all of which markedly, repeatedly and persistently disrupt the gut microbiome. Thus, this critical gap in the field needs to be addressed by a trial of FMT in SOT recipients with CDI.

ELIGIBILITY:
Inclusion Criteria:

* Is willing to provide written informed consent.
* Is willing to comply with all study procedures and be available for the duration of the study.
* Can take oral medication
* At least 18 years of age.
* Is a solid organ transplant (SOT) recipient
* Has had at recurrent C. difficile infection defined as: positive C. difficile testing in stool and diarrhea (three or more loose stools over 24 hours) during the 180 day period following completion of treatment for prior episode
* History of positive IgG test to cytomegalovirus (CMV) and Epstein-Barr Virus (EBV) for subject or donor
* Clinical response to 4-14 days of oral antibiotic standard of care treatment for the current episode of CDI. Clinical response is defined as greater than or equal to 25% reduction of diarrhea.
* Negative urine or serum pregnancy test for women of childbearing potential and agree to use effective form of contraception until 6 weeks post treatment

Exclusion Criteria:

* Major bowel resection surgery within 90 days of randomization
* Active intestinal disease (e.g. Crohn's disease, ulcerative colitis)
* History of total colectomy or bariatric surgery
* Known or suspected toxic megacolon and/or small bowel ileus
* Presence of colostomy or ileostomy.
* Taking concomitant antibiotics within 48 hours of Visit 2. Topical antibiotics, and antibiotics for transplant prophylaxis are permitted
* Dysphagia; oropharyngeal, S), or patient has evidence of dysphagia when the 'safety test' capsule is administered
* Currently receiving medication for treatment of acute rejection and/or develop acute rejection prior to administration of FMT
* Active, Severe Gastroparesis
* Unwilling to withhold probiotics. Probiotics include supplements, prescriptions, and non-prescriptions. Foods (like yogurt) are not prohibited
* Neutropenia, ≤ 500 neutrophils/ml [noted in medical records and resulted within 7 days of Visit 1])
* Symptomatic co-infection with another intestinal pathogen as determined by chart review
* Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for any active malignancy. Patients on maintenance chemotherapy could be enrolled after consultation with the study Medical Monitor
* Any severe food allergy, defined as a history of anaphylaxis, systemic urticarial or angioedema attributed to a food and requiring current avoidance precautions
* Expected life expectancy is less than 6 months
* Use of investigational drugs, biologics, or devices within 30 days prior to randomization.
* Women who are pregnant, lactating or planning on becoming pregnant during the study
* Not suitable for study participation due to other reasons at the discretion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - Mayo Clinic, Rochester, Minnesota
  - Ohio State University, Columbus, Ohio
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Pre-assignment Details: consent
Period: Overall Study
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Started | 0 | 3
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Low subject accrual
Groups:
- Total: Total of all reporting groups
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin | Total
Number analyzed (Participants) | 0 | 3 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 0 | 3 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Compare the Rate of Recurrence of CDI in Solid Organ Transplant Recipients With FMT Compared With Oral Vancomycin
Description: Recurrence is defined as diarrhea (greater or equal to 3 or more loose stools that take the shape of the collection container in a 24 hr period)
Time Frame: 60 consecutive days
Population: Target enrollment was not met and data cannot be compared as all enrolled subjects were randomized to 1 arm only.
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Number analyzed (Participants) | 0 | 3
Participants | 0 | 1

2. Secondary Outcome: CDI-related Quality of Life (QOL) Compared Using Treatment and Time Interaction as Model Terms While Adjusting for Potential Confounders
Description: Cdiff32 32-item questionnaire, with a range of 0 to 100, with 100 representing the best score, and 0 representing the worst score. Dietary component of the questionnaire linked to any stool microbiome data to determine whether diet influences gut microbiota.
Time Frame: Weeks 4, 29 weeks
Population: Study ended early per FDA-related COVID restrictions, samples not processed. No data available to report.
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Compare the Change in Gut Microbiota and Evaluate Changes in Microbiota to Assess for Safety of FMT in Patients
Description: Using multiple metric of microbiota structure and function, analyze gut microbiome samples to evaluate the association between change in gut microbiome and recurrent CDI
Time Frame: up to 30 weeks of study participation
Population: Study ended early per FDA-related COVID restrictions, samples not processed. No data available to report.
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Patients Who Experienced Short or Medium Term Adverse Events
Description: List and evaluate all short- and medium-term safety events as defined in the study protocol for the safety of FMT in SOT patients
Time Frame: Up 30 weeks of study participation
Population: Target enrollment was not reached and all subjects were randomized to 1 arm only, so planned analyses cannot be performed.
Measure: Count of Participants; unit: Participants
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Number analyzed (Participants) | 0 | 3
Participants | 0 | 1

5. Secondary Outcome: Compare the Effects of FMT and Oral Vancomycin on Intestinal Colonization by Multi-drug-resistant Organisms Other Than C. Difficile in SOT Patients
Description: Analysis all stool samples and compare the effects of FMT and oral vancomycin on intestinal colonization with multi-drug resistant organisms (other than C. difficile) in SOT patients
Time Frame: up to 30 weeks of study participation
Population: Study ended early per FDA-related COVID restrictions, samples not processed. No data available to report.
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 weeks
Description: No differences from standard definition of adverse events. Adverse events are inquired upon during weekly visits and follow-up phone visits by study staff.
Arm/Group | FMT Oral Capsules/ Oral Vancomycin Placebo | Placebo FMT Capsules/ Active Oral Vancomycin
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/0 | 1/3
Other Adverse Events (participants affected / at risk) | 0/0 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FMT Oral Capsules/ Oral Vancomycin Placebo (N=0) | Placebo FMT Capsules/ Active Oral Vancomycin (N=3)
Hospitalization due to toe infection (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/45/NCT03617445/Prot_SAP_005.pdf